CLINICAL TRIAL: NCT06966817
Title: The Effect of Two Different Oral Care Solutions on Ventilator-Associated Pneumonia and Oral Health of Mechanically Ventilated Patients in the Intensive Care Unit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AEŞH-EK1-2024-0034
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Ventilator-associated Pneumonia and Oral Health
Keywords: ventilator-associated pneumonia , oral health; ventilator-associated pneumonia ,oral health
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Before starting the study, the purpose of this study was explained to all nurses working in the intensive care unit and a 1-hour training was given about the study. The content of this training included theoretical information for nurses and guidance on the correct application of the oral care protocol. After the oral care application protocol in the intensive care unit was effectively implemented by the nurses, the data collection phase of the study was started.
  After the compliance of the patients admitted to the intensive care unit with the study inclusion criteria was evaluated, the oral care protocol to be applied to the patients was explained to the relatives of the patients included in the study and written and verbal consents were obtained.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Oral care for control group-1: First, the patient's teeth are brushed twice a day (06:00-18:00) with a small-headed, soft-bristled toothbrush, fluoride/non-foaming toothpaste and sterile water. Then, the mouth is aspirated to remove secretions and residues. After brushing, the sponge stick is dipped in 0.25% chlorhexidine solution and the mouth is cleaned in a way that it is used only once for each section of the mouth. In addition, between 12:00-24:00, the sponge stick is dipped in 0.25% chlorhexidine solution and the mouth is cleaned in a way that it is used only once for each section of the mouth.
  Interventions: Drug: control group(chlorhexidine)
- experimental group (Active Comparator): Oral care for experimental group-2: First, the patient's teeth are brushed twice a day (06:00-18:00) with a small-headed, soft-bristled toothbrush, fluoride/non-foaming toothpaste and sterile water. After brushing, the sponge swab is dipped into 0.05% cetylpyridinium chloride solution and the mouth is cared for in a way that it can be used only once for each part of the mouth. In addition, between 12:00 and 24:00, the sponge swab is dipped into 0.05% cetylpyridinium chloride solution and the mouth is cared for in a way that it can be used only once for each part of the mouth.
  Interventions: Drug: Experimental Group(cetylpyridinium chloride)

INTERVENTIONS:
Drug: control group(chlorhexidine) — The sponge swab is dipped in 0.25% chlorhexidine solution and used once for each part of the mouth, 4 times a day to provide oral care.
  Arms: control group
Drug: Experimental Group(cetylpyridinium chloride) — The mouth is cleaned by dipping a sponge swab into 0.05% cetylpyridinium chloride solution and using it once for each part of the mouth, 4 times a day.
  Arms: experimental group

SUMMARY:
The aim of this observational study is to evaluate the effects of two different oral care solutions on ventilator-associated pneumonia and oral health in mechanically ventilated participants in the intensive care unit.

Did oral health improve in participants who used cetylpyridinium chloride? Did pneumonia develop? Did oral health improve in participants who used chlorhexidine chloride? Did pneumonia develop? The results will be evaluated by giving oral care to the participants with these solutions for 5 days with the same protocol.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is defined as pulmonary parenchymal infection in patients exposed to invasive mechanical ventilation for at least 48 hours and is a part of intensive care unit (ICU)-acquired pneumonia. Ventilator-associated pneumonia is the most common intensive care unit (ICU)-acquired infection among patients receiving invasive mechanical ventilation. When the VAP data of surgical and medical ICUs of thirty-six developing countries, including our country, for the years 2013-2018 were evaluated; the average VAP rate was determined as 11.47 per 1000 ventilator days. It contributes to the increase in hospital mortality, MV and ICU hospital stay. Therefore, it worsens the condition of the critically ill patient and increases the total hospitalization cost. It has become mandatory to take preventive measures to ensure control and reduce the incidence of VAP. Preventive strategies to prevent the development of pneumonia in ventilated patients are based on the implementation of infection control, i.e., avoiding prolonged ventilation with adequate sedation and weaning protocols, avoiding biofilm formation on the endotracheal tube and microaspiration of subglottic secretions, avoiding bacterial translocation from the stomach to the upper airway, and avoiding oropharyngeal colonization. Lack of effective oral hygiene results in the development of dental plaque deposits on the teeth within 72 hours, which can be reservoirs for potential respiratory pathogens. Bacteria present in plaque serve as a reservoir for potential pathogens that can enter the respiratory tract. Because of this potential for infection, oral hygiene is important in patients receiving mechanical ventilation. Keeping a patient's mouth clean and disease-free (oral hygiene) can help prevent VAP. Mouthwashes have been recommended as a regular oral care because they can reduce costs and reduce plaque formation. The type, concentration, dose, and frequency of use of the rinse may also affect antibacterial efficacy. There remains uncertainty regarding the most effective protocols, including the types of personnel involved, frequency of oral care, whether antiseptics should be used, and if so, what type of antiseptic to use (e.g., chlorhexidine gluconate, sodium bicarbonate, hydrogen peroxide, cetylpyridinium chloride, povidone-iodine). Currently, the Centers for Disease Control and Prevention (CDC) recommends oral hygiene with 0.12% chlorhexidine (CHX) during the perioperative period of cardiac surgery, but there are no recommendations for its routine use in the prevention of nosocomial pneumonia in critically ill patients. Cetylpyridinium chloride (CPC) is a broad-spectrum antimicrobial agent that has been shown to be effective in reducing dental plaque and preventing gingivitis. Cetylpyridinium chloride 0.05% has been used as an alternative to reduce dental plaque and gingivitis in patients who develop mucosal irritation and stains due to CHX.

In light of all this information, oral care is one of the most important treatments for mechanically ventilated patients in the intensive care unit. It supports the treatment of intensive care patients and can prevent respiratory tract infections. For this reason, it is important to determine the effectiveness of oral care solutions used in patients and their effects on ventilator-associated pneumonia.

The aim of this study is to evaluate the effects of two different oral care solutions on ventilator-associated pneumonia and oral health of patients on mechanical ventilation in the intensive care unit.

H0: There is no difference between the development of VAP and oral health of patients on mechanical ventilation in the intensive care unit where 0.25% chlorhexidine gluconate is used in oral care and the development of VAP and oral health of patients on mechanical ventilation in the intensive care unit where 0.05% cetylpyridinium chloride is used in oral care.

H1: There is a difference between the development of VAP and oral health of patients on mechanical ventilation in the intensive care unit where 0.25% chlorhexidine gluconate is used in oral care and the development of VAP and oral health of patients on VAP and oral health of patients on oral care who 0.05% cetylpyridinium chloride is used in oral care.

ELIGIBILITY:
Inclusion Criteria:• Being 18 years of age or older

* Requiring mechanical ventilation for at least 48 hours
* Not having a diagnosis of aspiration pneumonia
* Having a Clinical Lung Infection Score (CPIS) <6 on the first day
* Not having a diagnosis of pneumonia or COVID
* Not having facial or oral trauma
* Being within the first 24 hours of the intubation process
* Not having a medical impediment to elevating the head of the bed 30o

Exclusion Criteria:

* Not accepting to participate in the study
* Termination of MV support for less than 48 hours
* Being allergic to any of the solutions to be used in oral care
* Being diagnosed with immunodeficiency
* Having thrombocytopenia, leukopenia and oral aphthae, stomatitis, candidiasis, gingivitis
* Using immunosuppressive drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
EFFECTS OF TWO DIFFERENT ORAL CARE SOLUTIONS ON VENTILATOR-ASSOCIATED PNEUMONIA AND ORAL HEALTH OF PATIENTS CONNECTED TO MECHANICAL VENTILATORS IN THE INTENSIVE CARE UNIT | from registration until the end of the 5th day
  The same person evaluates the patients' mouths every day at 07:00 with the oral hygiene oral assessment scale.
  On the 1st, 3rd and 5th days, patients are evaluated with the clinical pulmonary infection score. After all these evaluations, the patient is diagnosed with pneumonia or not by the intensive care specialist.

CONTACTS AND LOCATIONS:
Overall Officials: bediye öztaş, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided